CLINICAL TRIAL: NCT05445219
Title: Identifying Therapeutic Hemodialysis Targets Through Cerebrovascular Reactivity; RESPIRACT 2
Acronym: RESPIRACT 2
Status: Active, not recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Chris McIntyre, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 121136
Record Dates: First submitted 2022-06-27; First posted 2022-07-06 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Chronic Kidney Failure
Keywords: Hemodialysis; Cerebrovascular Reactivity; Cognitive Impairment
MeSH Terms: conditions — Kidney Failure, Chronic; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: RespirAct — The RespirAct device is an automated breathing circuit that uses a gas bladder to control and deliver CO2 to measure cerebrovascular reactivity

SUMMARY:
Patients with chronic kidney disease receiving hemodialysis (HD) suffer from higher rates of brain vascular disease and decreased cognition than the general population. One way to assess brain vascular health and response to HD stress, is to test how the brain's blood flow responds to carbon dioxide (CO2) to measure Cerebrovascular Reactivity (CVR). In this study, the investigators will compare the magnitude and speed of the brain's blood flow response to a step-wise change in CO2 with hemodynamic, dialysis, and cognitive parameters. The goal of the study is to establish therapeutic targets that can be altered during the dialysis procedure to protect the brain from HD stress.

DETAILED DESCRIPTION:
This is a follow-up study previously conducted by our lab group titled: "Hemodialysis Patients Have Impaired Cerebrovascular Reactivity to CO2 Compared to Chronic Kidney Disease Patients and Healthy Controls: A Pilot Study". It was determined that individuals who receive hemodialysis (HD) exhibited significant differences in their Cerebrovascular Reactivity (CVR) when compared to both healthy controls, and patients with kidney disease not yet on HD.

In this study, the aim is to determine if the degree of cognitive impairment is related to the degree of impaired brain blood flow response in order to determine therapeutic targets that may be altered during the dialysis procedure in order to preserve cognitive functioning in the patient's receiving HD, building upon the previous feasibility study.

This study will require 4 assessments over the course of 2 dialysis treatments (2 assessments per dialysis treatment [ie. pre and post HD assessments]). The subsequent dialysis treatment assessments will be completed in the course of a month to mitigate learning effects with regards to the cognitive assessment.

The study assessment includes:

1. Measuring cerebrovascular reactivity (CVR) before and after hemodialysis (HD):

   CVR will be measured using two specialized devices: RespirActTM in combination with Transcranial Doppler before and after an HD session. Specifically, the RespirActTM device is an automated breathing circuit that uses a gas bladder to control and deliver carbon dioxide (CO2). It has various gas cylinders that are used in order to obtain the correct increase in CO2 in each patient. This type of gas manipulation was selected because it is a more accurate measure of CVR, while also reducing between-subject variability.

   Transcranial Doppler is used in conjunction with the RespirActTM to allow insight into cerebral blood flow, by measuring the middle cerebral artery's blood flow velocity.

   During the CVR measurement, the RespirActTM will be connected to a facemask, and the Transcranial Doppler will be positioned on the trans-temporal window.

   During the diagnostic assessment there will be three steps:
   1. Baseline: Measurement of CVR and hemodynamics with no CO2 stimulus applied. Will take approximately 5 minutes.
   2. CO2 Diagnostic Assessment: Inducement of hypercapnia by raising baseline CO2 levels to 5-10 mmHg above baseline. This causes controlled stress, allowing insight into how the brain responds to stress. This increase will be sustained for approximately 5 minutes.
   3. Return to baseline: CO2 stimulus is removed and the patient is monitored until levels return to baseline. Will take roughly 5 minutes.

   Note: time intervals may be shortened or lengthened if the patient feels uncomfortable, asks to cease the application of CO2, or needs longer to return to baseline.
2. Identification of potential hemodynamic and dialysis targets:

   By investigating hemodynamic and specific HD parameters, identifiable targets may be ascertained that can be used to protect the brain during HD by investigating CVR before and after an HD session. To measure hemodynamic parameters the Finapres NOVA, a finger cuff device that allows for non-invasive real-time capture and recording of heart rate, blood pressure, and mean arterial pressure will be implemented. Blood samples will also be collected pre and post HD (done through the dialysis access point), which will give insight into potential dialysis targets such as sodium, calcium, magnesium, acid-base balance, and inflammation with respect to CVR.
3. Determining how CVR, cognitive impairment, and the HD process are related:

By performing a cognitive assessment before and after the HD treatment, it will allow insight into how the brain is affected by the HD process, along with how it is related to CVR. The cognitive assessment battery selected is as follows:

1. A web based cognitive assessment: The Cambridge Brain Sciences (CBS) is a computerized cognitive assessment that can be self-administered. The version that entails 6 tasks which primarily measure verbal ability, short term memory, and reasoning skills has been selected for this study. The CBS will be used in conjunction with a dementia screening tool Montreal Cognitive Assessment (MoCA), as earlier work demonstrated that CBS helps screening tools differentiate cognitive impairment while providing a more comprehensive insight into cognitive impairment, particularly with individuals who demonstrated borderline impairment.
2. A traditional screening tool: The MoCA is a quick dementia screening instrument that can detect mild cognitive impairment by assessing different cognitive domains, such as attention, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation, but still gives an overall assessment of global cognitive function. The MoCA has a maximum score of 30 with traditionally scores below 26 (1 standard deviation (SD)) indicating mild cognitive impairment (MCI), however a cut-off of 1.5SD for a measure of MCI, which has been derived from the diagnostic criteria from the Cardiovascular Health Cognition Study and the Mayo Clinic Study of Aging.
3. A commonly used attention and executive function assessment in those with kidney disease: The Trails Making Test (TMT) is composed of 2 subtests: TMTA and TMTB. In the TMTA the patient is asked to connect the numbers 1 through 25 as quickly as possible. It is a measure of visuomotor tracking, scanning, and attention. Alternatively, the TMTB adds an extra layer to the TMTA in that the patient is now asked to alternate numbers and letters (1-A-2-B-3-C etc.) which requires thinking flexibility and mental shifting and executive function.

In total this assessment should take 45 minutes to complete each time.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old, receiving hemodialysis treatment at least 3 times per week at a London Health Sciences Centre facility
* English proficiency

Exclusion Criteria:

* Mental incapacity to consent
* Declined to participate
* Severe chronic obstructive lung disease (COPD) /Asthma
* History of cerebrovascular accident (stroke, transient ischemic attack)
* Previous neurosurgery
* History of carotid stenosis or carotid surgery
* History of vasculitis
* Documented Dementia
* Pregnancy
* Not fluent in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 18 years old, receiving hemodialysis treatment at least 3 times per week at a London Health Sciences Centre facility
Sampling Method: Non-Probability Sample
Enrollment: 37 (Estimated)
Dates: Start 2023-05-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Baseline RespirAct measurement Pre Dialysis Weekday Treatment | 20 minutes to complete the assessment before HD treatment
  The CVR diagnostic assessment with the RespirAct will be performed prior to the dialysis treatment by all consenting patients on a weekday HD session. Examining CVR before the dialysis session will allow for insight into the patient's baseline CVR function. CVR via the RespirAct device is an automated breathing circuit that uses a gas bladder to control and deliver carbon dioxide (CO2). It has various gas cylinders that are used in order to obtain the correct increase in CO2 in each patient.
RespirAct measurement Post Dialysis Weekday Treatment | 20 minutes to complete the assessment after HD treatment
  The CVR diagnostic assessment with the RespirAct will be performed after the dialysis treatment by all consenting patients on a weekday HD session. Examining CVR after the dialysis session will allow for insight into how the patient's CVR function has been altered by the dialysis treatment. CVR via the RespirAct device is an automated breathing circuit that uses a gas bladder to control and deliver carbon dioxide (CO2). It has various gas cylinders that are used in order to obtain the correct increase in CO2 in each patient.
Baseline RespirAct measurement Pre Dialysis Weekend Treatment | 20 minutes to complete the assessment before HD treatment
  The CVR diagnostic assessment with the RespirAct will be performed prior to the dialysis treatment by all consenting patients on a weekend HD session. Examining CVR before the dialysis session will allow for insight into the patient's baseline CVR function. By timing this assessment after the weekend dialysis break insight into how CV is affected by fluid status can be observed. CVR via the RespirAct device is an automated breathing circuit that uses a gas bladder to control and deliver carbon dioxide (CO2). It has various gas cylinders that are used in order to obtain the correct increase in CO2 in each patient.
RespirAct measurement Post Dialysis Weekend Treatment | 20 minutes to complete the assessment after HD treatment
  The CVR diagnostic assessment with the RespirAct will be performed after the dialysis treatment by all consenting patients on a weekend HD session. Examining CVR after the dialysis session will allow for insight into how the patient's CVR function has been altered by the dialysis treatment. Specifically, HD sessions after the weekend dialysis break require higher ultrafiltration rates as more fluid is retained by the patients. This leads to a more aggressive treatment to get the patient down to their dry weight. Therefore, having this treatment follow the weekend break dialysis treatment the intensity of dialysis treatment and its effects on CVR can be assessed. CVR via the RespirAct device is an automated breathing circuit that uses a gas bladder to control and deliver carbon dioxide (CO2). It has various gas cylinders that are used in order to obtain the correct increase in CO2 in each patient.
Baseline Doppler measurement Pre Dialysis Weekday Treatment | 20 minutes to complete the assessment before HD treatment
  The CVR diagnostic assessment also needs to include Doppler in order to obtain arterial blood flow velocity. This will be performed prior to the dialysis treatment by all consenting patients on a weekday HD session. Examining CVR before the dialysis session will allow for insight into the patient's baseline CVR function.
Doppler measurement Post Dialysis Weekday Treatment | 20 minutes to complete the assessment before HD treatment
  The CVR diagnostic assessment also needs to include Doppler in order to obtain arterial blood flow velocity. This will be performed after the dialysis treatment by all consenting patients on a weekday HD session. Examining CVR after the dialysis session will allow for insight into whether the patient's CVR function was changed by the HD treatment.
Baseline Doppler measurement Pre Dialysis Weekend Treatment | 20 minutes to complete the assessment before HD treatment
  The CVR diagnostic assessment also needs to include Doppler in order to obtain arterial blood flow velocity. This will be performed prior to the dialysis treatment by all consenting patients on a weekday HD session. Examining CVR before the dialysis session will allow for insight into the patient's baseline CVR function while having more fluid retained, as there has been a weekend break since the last HD session.
Doppler measurement Post Dialysis Weekend Treatment | 20 minutes to complete the assessment after HD treatment
  The CVR diagnostic assessment also needs to include Doppler in order to obtain arterial blood flow velocity. This will be performed after the dialysis treatment by all consenting patients on a weekday HD session. Examining CVR after the dialysis session will allow for insight into whether the patient's CVR function was changed by the HD treatment. Having this treatment follow the weekend break dialysis treatment the intensity of dialysis treatment and its effects on CVR can be assessed.

SECONDARY OUTCOMES:
Heart Rate Monitoring by Finapres NOVA- weekday treatment | Duration of the CVR assessment and HD treatment (roughly 4.5 hours)
  Hemodynamic parameters will be investigated by the use of the Finapres NOVA which is a finger cuff device that allows for non-invasive real-time capture and recording of heart rate, blood pressure, and mean arterial pressure. Monitoring for the whole length of treatment and the CVR assessment will give insight into how hemodynamics change throughout the dialysis and CVR assessment.
Blood Pressure Monitoring by Finapres NOVA- weekday treatment | Duration of the CVR assessment and HD treatment (roughly 4.5 hours)
  Hemodynamic parameters will be investigated by the use of the Finapres NOVA which is a finger cuff device that allows for non-invasive real-time capture and recording of heart rate, blood pressure, and mean arterial pressure. Monitoring for the whole length of treatment and the CVR assessment will give insight into how hemodynamics change throughout the dialysis and CVR assessment.
Mean Arterial Pressure Monitoring by Finapres NOVA- weekday treatment | Duration of the CVR assessment and HD treatment (roughly 4.5 hours)
  Hemodynamic parameters will be investigated by the use of the Finapres NOVA which is a finger cuff device that allows for non-invasive real-time capture and recording of heart rate, blood pressure, and mean arterial pressure. Monitoring for the whole length of treatment and the CVR assessment will give insight into how hemodynamics change throughout the dialysis and CVR assessment.
Heart Rate Monitoring by Finapres NOVA- weekend treatment | Duration of the CVR assessment and HD treatment (roughly 4.5 hours)
  Hemodynamic parameters will be investigated by the use of the Finapres NOVA which is a finger cuff device that allows for non-invasive real-time capture and recording of heart rate, blood pressure, and mean arterial pressure. Monitoring for the whole length of treatment and the CVR assessment will give insight into how hemodynamics change throughout the dialysis and CVR assessment. Additionally, since this treatment is after the dialysis weekend break insight will be provided on how more aggressive dialysis treatments ( ex higher ultrafiltration rates) affect hemodynamic properties.
Blood Pressure Monitoring by Finapres NOVA- weekend treatment | Duration of the CVR assessment and HD treatment (roughly 4.5 hours)
  Hemodynamic parameters will be investigated by the use of the Finapres NOVA which is a finger cuff device that allows for non-invasive real-time capture and recording of heart rate, blood pressure, and mean arterial pressure. Monitoring for the whole length of treatment and the CVR assessment will give insight into how hemodynamics change throughout the dialysis and CVR assessment. Additionally, since this treatment is after the dialysis weekend break insight will be provided on how more aggressive dialysis treatments ( ex higher ultrafiltration rates) affect hemodynamic properties.
Mean Arterial Pressure Monitoring by Finapres NOVA- weekend treatment | Duration of the CVR assessment and HD treatment (roughly 4.5 hours)
  Hemodynamic parameters will be investigated by the use of the Finapres NOVA which is a finger cuff device that allows for non-invasive real-time capture and recording of heart rate, blood pressure, and mean arterial pressure. Monitoring for the whole length of treatment and the CVR assessment will give insight into how hemodynamics change throughout the dialysis and CVR assessment. Additionally, since this treatment is after the dialysis weekend break insight will be provided on how more aggressive dialysis treatments ( ex higher ultrafiltration rates) affect hemodynamic properties.
Blood Collection- Pre Dialysis Weekday Treatment | Less than a minute to complete the assessment before HD treatment
  Routine blood work will be collected via the patient's dialysis access point by the renal staff. The analysis will determine the hemodynamic status and kidney status of the patient before dialysis.
Blood Collection-Post Dialysis Weekday Treatment | Less than a minute to complete the assessment after HD treatment
  Routine blood work will be collected via the patient's dialysis access point by the renal staff. The analysis will determine the hemodynamic status and kidney status of the patient after dialysis.
Blood Collection-Pre Dialysis WeekendTreatment | Less than a minute to complete the assessment before HD treatment
  Routine blood work will be collected via the patient's dialysis access point by the renal staff. The analysis will determine the hemodynamic status and kidney status of the patient before dialysis.
Blood Collection-Post Dialysis Weekend Treatment | Less than a minute to complete the assessment after HD treatment
  Routine blood work will be collected via the patient's dialysis access point by the renal staff. The analysis will determine the hemodynamic status and kidney status of the patient after dialysis.
Cambridge Brain Sciences Pre Dialysis weekday assessment | Less than 10 minutes to complete the assessment before HD treatment
  Cambridge Brain Sciences (CBS) 6 task version measures verbal ability, short-term memory, and reasoning skills. It is a computerized assessment performed on a tablet. Pre-dialysis assessment will give insight into the cognitive baseline before dialysis and will be related to hemodynamics and CVR outcomes. Scores are determined by the time to complete and number of errors.
Cambridge Brain Sciences Pre Dialysis weekend assessment | Less than 10 minutes to complete the assessment before HD treatment
  Cambridge Brain Sciences (CBS) 6 task version measures verbal ability, short-term memory, and reasoning skills. It is a computerized assessment performed on a tablet. Pre-dialysis assessment will give insight into the cognitive baseline before dialysis and how it relates to the degree of fluid retention after the weekend dialysis break. Will be related to hemodynamics and CVR outcomes. Scores are determined by the time to complete and number of errors.
Cambridge Brain Sciences Post Dialysis weekday assessment | Less than 10 minutes to complete the assessment after HD treatment
  Cambridge Brain Sciences (CBS) 6 task version measures verbal ability, short-term memory, and reasoning skills. It is a computerized assessment performed on a tablet. Post dialysis assessment will give insight into how the cognitive status has changed after the HD treatment. Will be related to hemodynamics and CVR outcomes. Scores are determined by the time to complete and number of errors.
Cambridge Brain Sciences Post Dialysis weekend assessment | Less than 10 minutes to complete the assessment after HD treatment
  Cambridge Brain Sciences (CBS) 6 task version measures verbal ability, short-term memory, and reasoning skills. It is a computerized assessment performed on a tablet. Post dialysis assessment will give insight into how the cognitive status has changed after a more aggressive HD treatment following the weekend break. Will be related to hemodynamics and CVR outcomes. Scores are determined by the time to complete and number of errors.
Montreal Cognitive Assessment Pre Dialysis weekday assessment | Less than 5 minutes to complete the assessment before HD treatment
  The Montreal Cognitive Assessment (MoCA) is a quick dementia screening instrument that can detect mild cognitive impairment by assessing different cognitive domains, such as attention, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation, but still gives an overall assessment of global cognitive function. The MoCA has a maximum score of 30 with traditionally scores below 26 (1 standard deviation (SD)) indicating MCI, however, we will use a cut-off of 1.5SD for a measure of MCI, which has been derived from the diagnostic criteria from the Cardiovascular Health Cognition Study and the Mayo Clinic Study of Aging. Pre-dialysis assessment will give insight into the cognitive baseline before dialysis and will be related to hemodynamics and CVR outcomes.
Montreal Cognitive Assessment Pre Dialysis weekend assessment | Less than 5 minutes to complete the assessment before HD treatment
  The Montreal Cognitive Assessment (MoCA) is a quick dementia screening instrument that can detect mild cognitive impairment by assessing different cognitive domains, such as attention, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation, but still gives an overall assessment of global cognitive function. The MoCA has a maximum score of 30 with traditionally scores below 26 (1 standard deviation (SD)) indicating MCI, however, we will use a cut-off of 1.5SD for a measure of MCI, which has been derived from the diagnostic criteria from the Cardiovascular Health Cognition Study and the Mayo Clinic Study of Aging. Pre-dialysis assessment will give insight into the cognitive baseline before dialysis and how it relates to the degree of fluid retention after the weekend dialysis break. Will be related to hemodynamics and CVR outcomes.
Montreal Cognitive Assessment Post Dialysis weekday assessment | Less than 5 minutes to complete the assessment after HD treatment
  The Montreal Cognitive Assessment (MoCA) is a quick dementia screening instrument that can detect mild cognitive impairment by assessing different cognitive domains, such as attention, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation, but still gives an overall assessment of global cognitive function. The MoCA has a maximum score of 30 with traditionally scores below 26 (1 standard deviation (SD)) indicating MCI, however, we will use a cut-off of 1.5SD for a measure of MCI, which has been derived from the diagnostic criteria from the Cardiovascular Health Cognition Study and the Mayo Clinic Study of Aging. Post dialysis assessment will give insight into how the cognitive status has changed after the HD treatment. Will be related to hemodynamics and CVR outcomes.
Montreal Cognitive Assessment Post Dialysis weekend assessment | Less than 5 minutes to complete the assessment after HD treatment
  The Montreal Cognitive Assessment (MoCA) is a quick dementia screening instrument that can detect mild cognitive impairment by assessing different cognitive domains, such as attention, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation, but still gives an overall assessment of global cognitive function. The MoCA has a maximum score of 30 with traditionally scores below 26 (1 standard deviation (SD)) indicating MCI, however, we will use a cut-off of 1.5SD for a measure of MCI, which has been derived from the diagnostic criteria from the Cardiovascular Health Cognition Study and the Mayo Clinic Study of Aging. Post dialysis assessment will give insight into how the cognitive status has changed after a more aggressive HD treatment following the weekend break. Will be related to hemodynamics and CVR outcomes.
Trails Making Test A Pre Dialysis weekday assessment | Less than 1 minutes to complete the assessment before HD treatment
  In the Trails Making Test A (TMTA) the patient is asked to connect the numbers 1 through 25 as quickly as possible. It is a measure of visuomotor tracking, scanning, and attention. Pre-dialysis assessment will give insight into the cognitive baseline before dialysis and will be related to hemodynamics and CVR outcomes. Scores are determined by the time to complete with the average completion time by controls being 40 seconds.
Trails Making Test A Post Dialysis weekday assessment | Less than 1 minutes to complete the assessment after HD treatment
  In the Trails Making Test A (TMTA) the patient is asked to connect the numbers 1 through 25 as quickly as possible. It is a measure of visuomotor tracking, scanning, and attention. Scores are determined by the time to complete with the average completion time by controls being 40 seconds.Post dialysis assessment will give insight into how the cognitive status has changed after the HD treatment. Will be related to hemodynamics and CVR outcomes.
Trails Making Test A Pre Dialysis weekend assessment | Less than 1 minutes to complete the assessment before HD treatment
  In the Trails Making Test A (TMTA) the patient is asked to connect the numbers 1 through 25 as quickly as possible. It is a measure of visuomotor tracking, scanning, and attention. Scores are determined by the time to complete with the average completion time by controls being 40 seconds. Pre-dialysis assessment will give insight into the cognitive baseline before dialysis and how it relates to the degree of fluid retention after the weekend dialysis break. Will be related to hemodynamics and CVR outcomes.
Trails Making Test A Post Dialysis weekend assessment | Less than 1 minutes to complete the assessment after HD treatment
  In the Trails Making Test A (TMTA) the patient is asked to connect the numbers 1 through 25 as quickly as possible. It is a measure of visuomotor tracking, scanning, and attention. Scores are determined by the time to complete with the average completion time by controls being 40 seconds. Post dialysis assessment will give insight into how the cognitive status has changed after a more aggressive HD treatment following the weekend break. Will be related to hemodynamics and CVR outcomes.
Trails Making Test B Pre Dialysis weekday assessment | Less than 2 minutes to complete the assessment before HD treatment
  The Trails Making Test B (TMTB) adds an extra layer to the TMTA in that the patient is now asked to alternate numbers and letters (1-A-2-B-3-C etc.) which requires thinking flexibility and mental shifting and executive function. Pre-dialysis assessment will give insight into the cognitive baseline before dialysis and will be related to hemodynamics and CVR outcomes. Scores are determined by the time to complete with the average completion time by controls being 94 seconds.
Trails Making Test B Post Dialysis weekday assessment | Less than 2 minutes to complete the assessment after HD treatment
  The Trails Making Test B (TMTB) adds an extra layer to the TMTA in that the patient is now asked to alternate numbers and letters (1-A-2-B-3-C etc.) which requires thinking flexibility and mental shifting and executive function. Scores are determined by the time to complete with the average completion time by controls being 94 seconds. Post dialysis assessment will give insight into how the cognitive status has changed after the HD treatment. Will be related to hemodynamics and CVR outcomes.
Trails Making Test B Pre Dialysis weekend assessment | Less than 2 minutes to complete the assessment before HD treatment
  The Trails Making Test B (TMTB) adds an extra layer to the TMTA in that the patient is now asked to alternate numbers and letters (1-A-2-B-3-C etc.) which requires thinking flexibility and mental shifting and executive function. Scores are determined by the time to complete with the average completion time by controls being 94 seconds. Pre-dialysis assessment will give insight into the cognitive baseline before dialysis and how it relates to the degree of fluid retention after the weekend dialysis break. Will be related to hemodynamics and CVR outcomes.
Trails Making Test B Post Dialysis weekend assessment | Less than 2 minutes to complete the assessment after HD treatment
  The Trails Making Test B (TMTB) adds an extra layer to the TMTA in that the patient is now asked to alternate numbers and letters (1-A-2-B-3-C etc.) which requires thinking flexibility and mental shifting and executive function. Scores are determined by the time to complete with the average completion time by controls being 94 seconds. Post dialysis assessment will give insight into how the cognitive status has changed after a more aggressive HD treatment following the weekend break. Will be related to hemodynamics and CVR outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher W McIntyre, MD/PHD, Principal Investigator — London Health Sciences Centre - Victoria Hospital
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No